CLINICAL TRIAL: NCT04770233
Title: Improving the Treatment of Anterior Cruciate Ligament Tears in Norway With Register-RCTs - Who Should Have Surgery
Brief Title: How to Best Treat Anterior Cruciate Ligament Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Norwegian National Knee Ligament Registry (Unknown); Sorlandet Hospital HF (Other Government); Kristiansund Hospital (Other); Asker & Baerum Hospital (Other)
Responsible Party: Principal Investigator, Guri Ranum Ekås, Consultant, Orthopedic Surgeon, Researcher, Assistant professor (MD/PhD), University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC148805
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: acl; anterior cruciate ligament injury; anterior cruciate ligament rupture; anterior cruciate ligament tear; secondary meniscal tear; ACL reconstruction; ACL rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Registry-based multi-center RCT. Centralized randomization through NNKLR stratified by participating centers. Allocation concealment secured by requiring registration into the NNKLR and the R-RCT before allocation is revealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early ACL reconstruction (Active Comparator): Early ACL reconstruction is performed within 12 weeks after ACL injury and is followed by rehabilitation led by a physiotherapist. ACL surgical technique and rehabilitation is pragmatic according to the routines at the including centre.
  Interventions: Procedure: Early ACL reconstruction
- Primary ACL rehabilitation (Active Comparator): Primary ACL rehabilitation is active rehabilitaion led by a physiotherapist. Active rehabilitation will begin as early as possible after the ACL injury. The goal of rehabilitation is to stabilized the knee without an operation.
  ACL reconstruciton is still an option after 6 months if the knee is unstable or do not allow adequat return to physical activity. If the patient sustain new knee injuries secondary to the ACL injury or has major instability, ACL reconstruction may be necessary before 6 months. The patients randomized to active rehabilitation will be routinely followed-up at his/her local hospital at 6 months.
  Interventions: Procedure: Active rehabilitation

INTERVENTIONS:
Procedure: Early ACL reconstruction — ACL reconstruction followed by rehabilitation
  Other Names: ACL surgery
  Arms: Early ACL reconstruction
Procedure: Active rehabilitation — Non-operative treatment with active rehabilitation led by a physiotherapist with optional delayed surgery if indicated.
  Other Names: Non-operative treatment, physiotherapy, physical therapy
  Arms: Primary ACL rehabilitation

SUMMARY:
The project is a pragmatic registry-based RCT aiming to investigate ACL injury treatment. Study results will help fill knowledge gaps, facilitate shared decision making and strengthen patient treatment.

Included patients will be randomized to (1) early ACL surgery followed by rehabilitation or (2) active rehabilitation with optional delayed surgery if indicated.

Randomization and data collection is conducted through the Norwegian National Knee Ligament Registry (NNKLR) which is a well established population based ACL registry. Participation is based on informed consent to participate in the NNKLR and the registry-based RCT. The study uses the platform and outcome measures of the NNKLR to collect and measure data. The data will be stored as usual in the NNKLR, but RCT specific data will be exported for analysis and stored inTjenester for sensitive data (TSD). Data collected in NNKLR are: patient data (age, height, weight, activity level, smoking-and snuff habits), knee injury data (injury data, injury mechanism, additional knee injury), treatment (non-operative or ACL reconstruction, reoperation), surgical details (operation date, antibiotics, anti-coagulants, graft type and size, approach for femoral tunnel, additional injury and additional surgical procedure) and patient reported knee function at baseline, 2, 5 and 10 years. Also, x-rays and MRIs will be imported for included patients and stored in TSD.

DETAILED DESCRIPTION:
Despite years of research on treating ACL injuries, it remains uncertain who should undergo reconstructive surgery and who should not.

Our project aims to provide definitive answers to these important clinical questions affecting more than 4,000 patients each year in Norway. We will provide this information by conducting a large comparative effectiveness trial of standard treatments for ACL deficiency. This RCT exploit the infrastructure of the Norwegian National Knee Ligament Registry (NNKLR), which uniquely include non-surgically treated ACL-tears and has almost complete coverage of surgical reconstructions. Our multi-center register-RCT design considerably reduces costs and enables us to more rapidly include many more patients. Consequently, the design and study size will give the results excellent external validity.

Surgery or not? It is estimated that 50% of patients with an ACL tear are treated surgically with a reconstruction.[1, 2] The majority of patients are young and active.[3] The general consensus in Scandinavia is that patients who manage to regain acceptable knee function after active rehabilitation alone should not initially have surgery. This treatment algorithm is supported mainly by only one high-quality randomized controlled trial.[4, 5] Prospective studies have reported that the functional recovery, the long term patient outcome and the radiographic sign of osteoarthritis are similar between patients treated surgically or non-surgically.[6-8] However, conclusion about cause and effect cannot be made due to the study designs. A recent Cochrane review concluded that there is a low-quality evidence that there was no difference between surgical and non-surgical treatment, and studies with high external validity is lacking.[9] In the debate of early surgery or not, the risk of subsequent meniscal and chondral injury in an unstable knee is often highlighted by promoters for early surgery. However, the studies behind this argument reports on the correlation between the timing of surgery and concomitant meniscal and cartilage injuries rather than on whether the initial treatment chosen was surgical or non-surgical.[10] This introduces a selection bias as a patients having surgery late may not be representative of all non-surgically treated patients. The findings in a systematic review on this topic by authors in the project group high-light that the uncertain estimate of new meniscal tears after ACL injury should not guide clinical practice for all patients.[11] Even though joint stability often is achieved with surgery, the rate of return to pre-injury activity level after surgery is reported less than 50%, and no consistent results in reduction of the risk of later osteoarthritis have been shown.[12] Admittedly, the risk of serious complications after ACL reconstruction is in general low, however still potentially devastating to the knee function.[13, 14]

About the Norwegian National Knee Ligament Register

The NNKLR was established in 2004 as the world´s first national cruciate ligament register[15]. The NNKLR assesses the outcome based on the Knee Injury and Osteoarthritis Outcome Score (KOOS) which is the gold standard validated patient reported outcome measure (PROM) [16] and by recording revision surgeries or other surgeries to the index knee. Since 2004 cruciate ligament reconstructions performed in Norway have been reported to the register with subsequent registration of revision surgeries and with input of PROM at 2, 5 and 10 years postoperatively. Just below 3000 patients are included yearly in the register. This has provided a unique resource for research and quality assessment, detecting inferior surgical procedures and providing prognostic information to guide practice.[17] Registries have had two major weaknesses limiting overall research impact:

1. Non-operatively treated injuries have not been included. This selection bias severely skews the evidence base for treatment guidelines.[17, 18,19] The NNKLR has recently piloted a project trying to mend this weakness.[20] The license for NNKLR issued by the Norwegian Data Inspectorate has been amended to allow for inclusion of patient at the time of ACL injury, allowing for follow-up within the register for the patients not undergoing surgery.
2. The design is fundamentally that of a prospective cohort. This does not allow researchers to make firm conclusions about differences in outcome between treatments. This major weakness of all national ACL registers is due to the inherent bias of being mainly observational.

Register-RCT The classic RCT remedies confounding bias by randomly allocating patients to each treatment ensuring equal distribution of measured and, importantly, unmeasured characteristics. However, RCTs often have strict inclusion and exclusion criteria leading to diminished generalizability to the general population. One may ask what good are RCTs if they can answer questions regarding only a tiny fraction of the population.[21] They are often expensive and time-consuming, limiting the possible amount of patients included. Recently, as an answer to these limitations, the implementation of randomization into registers has been proposed, and termed "the register-based RCT" (R-RCT).[22] The promise of this approach has been highlighted in high-ranking journals as the "next disruptive technology in clinical research".[21] Simply put, patients are included in a quality register, and the treatment is randomized. The outcome data is collected automatically through the register, cutting the costs and simplifying the follow-up. Analysis of the subsequent register data can conclude on effect estimates between treatments with the same level of evidence as those from regular RCTs, only with a greater external validity. The feasibility R-RCTs has been shown mainly in trials relating to interventions in cardiology and has only very recently been used in orthopedic trauma surgery[23-25].

Recruitment problems has been highlighted as a challenge in a previous RCT on ACL treatment.[26] The R-RCT mediates this by facilitating multi-center collaboration to ensure rapid inclusion of patients in the proposed trials.

Hypotheses, aims and objectives The overall aim of this project is to assess the effect of surgical treatment and non-surgical treatment of patients with a complete tear of the anterior cruciate ligament as assessed with the KOOS which is the commonly accepted gold standard patient reported outcome measure for knee injuries [16].

Primary objectives Investigate the outcome of surgical and non-surgical treatment of ACL-injury through a multi-center register-based RCT with outcome collection of primary endpoints solely performed by the NNKLR

Project methodology The NNKLR follows the patients until 10 years and this is the minimum time the project will follow the included patients. We include in the consent the possibility to contact all patients after the regular follow-up by the NNKLR as we plan to follow-up patients until 20 years after the injury and we also include in the consent the possibility of linking to for example the Norwegian Arthroplasty Register.

Project arrangements, method selection and analyses All participating centers already care for patients with cruciate ligament injuries and have all necessary equipment for this. The data collection at inclusion will be solely through a secure web-based system (Medisinsk Registreringssystem (MRS)- Helse Midt-Norge IT). During the planning and running of the trial the research group will work closely with the NNKLR.

Methods The NNKLR is a national quality registry. Reporting surgically treated patients to the register is mandatory for the surgeon. The surgeon report patient-specific data and surgical details on either a paper form or through a secure web-based interface at the time of inclusion. Information on implants used at surgery is registered with stickers provided by the manufacturers attached on the paper form, and by scanning the barcodes providing the same information when reporting electronically. Identical patient-specific data is collected at inclusion for the patients treated non-surgically. The web-based interface is maintained by the Medical Register System in the IT department of Central Norway Regional Health Authority. The NNKLR will be the main source of outcome collection in the planned trials. The patient reports PROMs at the time of inclusion and at 2-, -5- and -10-year follow-up, either through a paper-form or electronically. Clinical follow-up with subsequent primary or revision ACL reconstructions or other knee surgery to the index or contralateral knee are to be reported to the register by the surgeon.

Study design The study design is a register-based multi-center RCT. The structured rehabilitation will be identical in both groups and follow standardized goal-oriented guidelines.[27, 28] Randomization strategy: Randomization will be performed when the patients are included at first visit through the NNKLR embedded randomization module developed and implemented in this project. We will utilize centralized randomization stratified by participating centers[29, 30] Allocation concealment will be secured by requiring registration into the NNKLR and the R-RCT before allocation is revealed.

Sample size calculation: The sample size calculation will be based on a standard deviation of 20 for KOOS Quality of Life, a 90 % statistical power to detect a minimally clinically relevant difference of 10 between the treatment groups, an alpha level of 0.05 and allowing for a 20% drop-out rate.[5] In the non-surgically vs. surgical treatment RCT without stratification for age and activity level this will require at least 230 patients. Allowing for sub-group analysis on activity levels based on best estimates will increase sample-size to approximately 328 patients.

Statistical analyses: All subjects randomized will be included in the analysis. Investigation of the primary endpoint will be performed using analysis of covariance for the different treatment groups, stratified by site and adjusted and unadjusted for baseline KOOS-scores.[31] Both intention-to-treat and as-treated analyses will be performed. An absence of a clinically relevant difference will be assumed if the confidence interval of the difference includes differences of less than 10 units between groups. Secondary endpoints will be analyzed by analysis of covariance (KOOS) and chi-square tests (return to pre-injury activity level). Additional data collected outside NNKLR is clinical imaging (MRI/x-rays) taken in the course of treatment. Resource use (health economy) will be analysed through linkage to other registers (eg. NPR, IPLOS, Reseptregister) as stated in the consent and if needed supplemented with data from the electronic patient record.

Funding The project is fully funded through Program for klinisk behandlingsforskning (KLINBEFORSK) with a grant for the period of 2020 through 2024. There are no financial interests involved for neither the researchers nor the patients in this RCT.

User involvement We have teamed up with a named user.

Ethical considerations and data handling All participants must give written informed consent to be included into both the NNKLR an the register-based RCT. The NNKLR has a standing license from the Norwegian Data Protection Authority ref.nr. 16/01130-3/CDG covering both non-operatively treated and surgically treated patients included in the registry. The protocol for the register-based RCT and user-approved consent have been reviewed and approved the Regional Committees on Medical and Health Research Ethics (REC SØ).Before patient inclusion, the Ethical Boards at the including centres will need to review and approve the protocol (currently approved at Akerhus University Hospital).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have sustained an acute ACL injury (must be possible to perform the "early surgery" treatment option within 12 weeks)
* Age 16-50 years and skeletally mature
* No previous surgery in the index knee or knee injury which influences rehabilitation
* Patient capable to undergo both surgery and rehabilitation

Exclusion Criteria:

• Elite athletes (Tegner 10) in pivoting sports and patients with additional knee injuries warranting repair

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 328 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
The mean change in the score for Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales: Knee Related Quality of Life and Sports and Recreational Function from baseline to 2, 5 and 10 years after inclusion | at the time of inclusion/surgery, 2 years, 5 years and 10 years
  Knee Injury and Osteoarthritis Outcome Score (KOOS) is a gold standard for patient reported outcome measures for knee injuries and knee osteoarthrities. This score has five subscales: pain, symptoms, function in daily living, function in sports and recreation and quality of life. Each subscale is calculated separately from 0-100. A score of 100 represent the best score possible, indicating no symptoms and a score of 0 is the worst possible score indicating extreme symptoms.

SECONDARY OUTCOMES:
Rate of new meniscal injuries | 1 year, 2 years, 5 years, 10 years
  We want to detect the rate of new meniscal injuries (in the index knee) in the study arm populations.
Rate of subsequent knee surgery to the index knee | 2, 5 and 10 years
  We want to detect the rate and type of resurgeries to the study arm populations e.g. meniscal surgery, revision ACL surgery, debridement due to infection
Mean change in additional KOOS-subscales from baseline to follow-up | 2, 5 and 10 years
  We want to detect mean changes in the subscales Pain, Symptoms and Activities of daily living. Each subscale is calculated separately from 0-100. A score of 100 represent the best score possible, indicating no symptoms and a score of 0 is the worst possible score indicating extreme symptoms.
Rate of subsequent treatment of an ACL-tear of the contralateral knee | 2, 5 and 10 years
  We want to detect the rate of new ACL injuries and treatment to the other knee.
Rate of return to preinjury activity level | 2, 5 and 10 years
  We want to detect the rate of patients returning to preinjury activity level after ACL injury. Activity level is based on al Hefti's scale 1-4 according to degree of pivoting. Level 1 is pivoting sport such as soccer, basket ball, team handball, floorball, rugby. Level 2 is sports with some pivoting such as tennis, squash, alpine skiing, twin tip skiing, martial arts, dancing. Level 3 is sports without pivoting such as cycling, running, strength training, swimming, spinning, cross-country skiing. Level 4 is no sports activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rune Jakobsen, PhD/MD, Study Chair — Akershus University Hospital, University of Oslo
Locations (2):
- Norway (2):
  - Orthopedic Department, Akershus University Hospital, Lørenskog, Akershus
  - Orthopedic division, Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ytterstad K, Granan LP, Engebretsen L. [The Norwegian Cruciate Ligament Registry has a high degree of completeness]. Tidsskr Nor Laegeforen. 2011 Feb 4;131(3):248-50. doi: 10.4045/tidsskr.10.0536. Norwegian. PMID 21304574
- [Background] Spindler KP, Wright RW. Clinical practice. Anterior cruciate ligament tear. N Engl J Med. 2008 Nov 13;359(20):2135-42. doi: 10.1056/NEJMcp0804745. No abstract available. PMID 19005197
- [Background] Granan LP, Engebretsen L, Bahr R. [Surgery for anterior cruciate ligament injuries in Norway]. Tidsskr Nor Laegeforen. 2004 Apr 1;124(7):928-30. Norwegian. PMID 15060639
- [Background] Ingelsrud LH, Terwee CB, Terluin B, Granan LP, Engebretsen L, Mills KAG, Roos EM. Meaningful Change Scores in the Knee Injury and Osteoarthritis Outcome Score in Patients Undergoing Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2018 Apr;46(5):1120-1128. doi: 10.1177/0363546518759543. Epub 2018 Mar 8. PMID 29517924
- [Background] Engebretsen L, Forssblad M, Lind M. Why registries analysing cruciate ligament surgery are important. Br J Sports Med. 2015 May;49(10):636-8. doi: 10.1136/bjsports-2014-094484. Epub 2015 Feb 2. No abstract available. PMID 25807159
- [Background] Seil R, Mouton C, Theisen D. How to get a better picture of the ACL injury problem? A call to systematically include conservatively managed patients in ACL registries. Br J Sports Med. 2016 Jul;50(13):771-2. doi: 10.1136/bjsports-2015-095027. Epub 2015 Sep 23. No abstract available. PMID 26400957
- [Background] Krumholz HM. Registries and selection bias: the need for accountability. Circ Cardiovasc Qual Outcomes. 2009 Nov;2(6):517-8. doi: 10.1161/CIRCOUTCOMES.109.916601. No abstract available. PMID 20031886
- [Background] Ekas GR, Engebretsen L. [The cruciate ligament register--due for a change?]. Tidsskr Nor Laegeforen. 2016 Feb 23;136(4):298. doi: 10.4045/tidsskr.15.1291. eCollection 2016 Feb 23. No abstract available. Norwegian. PMID 26905841
- [Background] Lauer MS, D'Agostino RB Sr. The randomized registry trial--the next disruptive technology in clinical research? N Engl J Med. 2013 Oct 24;369(17):1579-81. doi: 10.1056/NEJMp1310102. Epub 2013 Aug 31. No abstract available. PMID 23991657
- [Background] Mathes T, Buehn S, Prengel P, Pieper D. Registry-based randomized controlled trials merged the strength of randomized controlled trails and observational studies and give rise to more pragmatic trials. J Clin Epidemiol. 2018 Jan;93:120-127. doi: 10.1016/j.jclinepi.2017.09.017. Epub 2017 Sep 22. PMID 28951111
- [Background] Sims AL, Parsons N, Achten J, Griffin XL, Costa ML, Reed MR; CORNET trainee collaborative. A randomized controlled trial comparing the Thompson hemiarthroplasty with the Exeter polished tapered stem and Unitrax modular head in the treatment of displaced intracapsular fractures of the hip: the WHiTE 3: HEMI Trial. Bone Joint J. 2018 Mar 1;100-B(3):352-360. doi: 10.1302/0301-620X.100B3.BJJ-2017-0872.R2. PMID 29589786
- [Background] Yndigegn T, Hofmann R, Jernberg T, Gale CP. Registry-based randomised clinical trial: efficient evaluation of generic pharmacotherapies in the contemporary era. Heart. 2018 Oct;104(19):1562-1567. doi: 10.1136/heartjnl-2017-312322. Epub 2018 Apr 17. PMID 29666176
- [Background] Frobert O, Lagerqvist B, Olivecrona GK, Omerovic E, Gudnason T, Maeng M, Aasa M, Angeras O, Calais F, Danielewicz M, Erlinge D, Hellsten L, Jensen U, Johansson AC, Karegren A, Nilsson J, Robertson L, Sandhall L, Sjogren I, Ostlund O, Harnek J, James SK; TASTE Trial. Thrombus aspiration during ST-segment elevation myocardial infarction. N Engl J Med. 2013 Oct 24;369(17):1587-97. doi: 10.1056/NEJMoa1308789. Epub 2013 Aug 31. PMID 23991656
- [Background] Frobell RB, Lohmander LS, Roos EM. The challenge of recruiting patients with anterior cruciate ligament injury of the knee into a randomized clinical trial comparing surgical and non-surgical treatment. Contemp Clin Trials. 2007 May;28(3):295-302. doi: 10.1016/j.cct.2006.10.002. Epub 2006 Oct 6. PMID 17137844
- [Background] Eitzen I, Holm I, Risberg MA. Preoperative quadriceps strength is a significant predictor of knee function two years after anterior cruciate ligament reconstruction. Br J Sports Med. 2009 May;43(5):371-6. doi: 10.1136/bjsm.2008.057059. Epub 2009 Feb 17. PMID 19224907
- [Background] Pandis N. Randomization. Part 2: Minimization. Am J Orthod Dentofacial Orthop. 2011 Dec;140(6):902-4. doi: 10.1016/j.ajodo.2011.08.016. No abstract available. PMID 22133958
- [Background] FAITH Investigators. Fixation using alternative implants for the treatment of hip fractures (FAITH): design and rationale for a multi-centre randomized trial comparing sliding hip screws and cancellous screws on revision surgery rates and quality of life in the treatment of femoral neck fractures. BMC Musculoskelet Disord. 2014 Jun 26;15:219. doi: 10.1186/1471-2474-15-219. PMID 24965132
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558